CLINICAL TRIAL: NCT03640520
Title: Randomized Controlled Trial (RCT) to Evaluate the Impact of Online Training Tools Related to Pediatric Resuscitation in General EDs
Brief Title: Evaluation of Online Training Tools in Pediatric Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 17-014752
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Family-centered Care in Pediatric Resuscitation

STUDY DESIGN:
Intervention Model Description: Investigators will conduct an RCT of the FACETS online skills training module (intervention) vs. an online training module reviewing pediatric readiness standards for all EDs (control).
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants on each team at each site will be blinded as to treatment condition and to the study goal of evaluating family centered care. Study staff who rate team performance of FCC from videotaped simulated pediatric resuscitations will also be blinded as to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Family-centered & Trauma-informed Support in Pediatric Resuscitation (FACETS: Pediatric Resuscitation) is an online skills training module for health care professionals involved in pediatric resuscitation in general EDs. The module combines didactic information and scenario-based learning with opportunities for the learner to practice applying their knowledge of Family Centered Care (FCC) practices at key choice points in realistic pediatric resuscitation case scenarios. Training content is guided by evidence regarding FCC practices that are effective in reducing concurrent and ongoing emotional distress in children and family members, and in promoting child and family involvement and satisfaction with care.
  Interventions: Other: FACETS: Pediatric Resuscitation
- Control (Active Comparator): An online training module in which participants will receive information and policy education about national pediatric readiness standards for all EDs, including a brief mention of FCC as one of these standards, with no specific skills training in FCC. The module provides practice-relevant knowledge related to pediatric differences and pediatric readiness.
  Interventions: Other: Control

INTERVENTIONS:
Other: FACETS: Pediatric Resuscitation — Family-centered & Trauma-informed Support in Pediatric Resuscitation (FACETS: Pediatric Resuscitation) is an online skills training module for health care professionals involved in pediatric resuscitation in general EDs. The module combines didactic information and scenario-based learning with opportunities for the learner to practice applying their knowledge of FCC practices at key choice points in realistic pediatric resuscitation case scenarios. Training content is guided by evidence regarding FCC practices that are effective in reducing concurrent and ongoing emotional distress in children and family members, and in promoting child and family involvement and satisfaction with care.
  Arms: Intervention
Other: Control — An online training module in which participants will receive information and policy education about national pediatric readiness standards for all EDs (including a brief mention of family-centered care as one of these standards), with no specific skills training in FCC. The module provides practice-relevant knowledge related to pediatric differences and pediatric readiness
  Arms: Control

SUMMARY:
The primary objective is to conduct a randomized controlled trial (RCT) to assess the impact of an online skills training module on 1) individual providers' self-rated confidence and comfort with and current practice of family centered care (FCC) skills; and 2) assess team performance of FCC and resuscitative care skills during simulated pediatric resuscitation scenarios.

DETAILED DESCRIPTION:
Context: Each year, more than 30 million children are evaluated at >5,000 US Emergency Departments (EDs); more than 85% present to general EDs. Pediatric resuscitation is particularly high-stakes aspect of emergency care for which non-pediatric-specialized EDs are often unprepared. Evidence shows differential outcomes as well, including a difference in mortality in pediatric resuscitation between general EDs (40%) and pediatric EDs (22%). The toll goes beyond physical health outcomes - about 1 in 6 seriously ill children (and their parents) will go on to have persistent posttraumatic stress symptoms related to their medical condition and treatment experiences.

BACKGROUND AND RATIONALE:

This research is part of a larger project to create and disseminate the "Self-Assessment through Video Evaluation for Performance improvement in Emergency Department-based Pediatric Resuscitation" (SAVE PEDS) Toolkit. This web-based resource will enable general emergency departments (EDs) across the US to reliably self-assess, measure and iteratively improve their performance in pediatric resuscitation via video review, assessment and debriefing of simulated or actual patient care emergencies, and accessible training materials. The current trial will test an online skills training module intended to be delivered as part of SAVE PEDS. Aimed at healthcare professionals, the Family-centered & Trauma-informed Support in Pediatric Resuscitation (FACETS: Pediatric Resuscitation) training combines didactic information and scenario-based learning with opportunities for the learner to practice applying his/her knowledge at key choice points in realistic pediatric resuscitation scenarios.

Medical resuscitation is a high-stakes, fast-moving environment in which a variable team of health care professionals and ancillary staff must work together seamlessly to maximize patient outcomes. Pediatric resuscitation is a relatively rare occurrence across all emergency care, and especially true in the general hospital where providers may have less comfort and experience with the care of children, and hospitals have fewer pediatric-specific resources. Yet the general hospital, where 85% of children are seen for emergency care, must be constantly ready for the resuscitation of a critically ill/injured child.

Gaps are known to exist in accessibility of pediatric resuscitation equipment, resuscitation skill performance and guideline adherence. The reported difference in mortality in pediatric resuscitation between general (40%) and pediatric (22%) EDs may be directly related to these gaps. Significant gaps also exist in the delivery of family-centered care (FCC) in the ED. FCC has been defined as care that emphasizes respect for patient and family perspectives regarding health care, and encouragement of patient and family participation in care and decision-making. Only half of general EDs report having FCC policies for children. FCC can be a particular challenge in the resuscitation setting, with many competing priorities for the medical team's attention and focus.

For patients and families, pediatric resuscitation is an extremely stressful experience. Symptoms of posttraumatic stress disorder (PTSD) are common in children (and family) in the aftermath of pediatric critical illness and injury, and these symptoms have been associated with medication non-adherence, lower quality of life and poorer functional outcomes. There is strong support for the positive impact of family presence and family involvement in care / decision-making - on patient safety, patient and family satisfaction, and child and family emotional health. Meaningful implementation of FCC during resuscitation requires a set of skills for which few ED providers have had systematic training. Providers in general EDs have even fewer opportunities to learn or practice these skills as they relate to pediatric resuscitation.

Study Design: this is a multi-site RCT

Setting/Participants include a total of 6-8 general EDs - in community or non-pediatric-specialized hospitals - will participate. Within each ED, Investigators will enroll individual health care professionals who are involved in pediatric resuscitation in the ED.

Study Interventions and Measures:

Investigators will gather information on site level factors relative to hospital resources and ED volumes to categorize and describe EDs.

Participants will complete demographics and pre-survey assessing self-rated confidence and practice of FCC and pediatric resuscitation. 2-3 teams at each site will then participate in two simulated pediatric resuscitation scenarios incorporating family presence. At Intervention group sites, participants will then complete the online FCC training. At Control group sites, participants will complete an online training on national pediatric readiness standards for EDs. Teams will then complete two additional simulated scenarios, after which a debriefing session will be held. Participants not present for the simulation sessions will complete the intervention or control training online. Afterwards, participants will complete a post-survey assessing self-rated confidence and practice of FCC and pediatric resuscitation. Four to twelve weeks post-training, teams at each site will participate in two additional simulation scenarios incorporating family presence.

STUDY OBJECTIVES

This randomized controlled trial (RCT) will be conducted in general ED settings, to evaluate the impact of the FACETS: Pediatric Resuscitation training module on:

1. individual providers' confidence and use of FCC skills in pediatric resuscitation (primary objective)
2. team performance of FCC and resuscitative care skills during simulated pediatric resuscitations (secondary objective).

STUDY PLAN

Investigators will conduct an RCT of the FACETS online training module (intervention) vs. an online training module reviewing pediatric readiness standards for all EDs (control) in six to eight participating institutions that are general non-pediatric-specialized EDs.

Randomization of the participating EDs will occur at the site level, with half allocated to the intervention condition and half to the control condition. All participants will be blinded as to treatment condition and as to the specific study goal of evaluating FCC. Study staff who rate team performance from videotaped simulated pediatric resuscitations will be blinded as to study condition.

Within each institution, Investigators will enroll individual health care professionals who are involved in pediatric resuscitation in the ED. An email invitation to all eligible staff will include a link to study consent and to the study pre-survey, both administered via REDCap.

All participants will complete the pre-training survey, either the intervention or the control training module, and the post-training survey. A subset of participants (based on availability) will additionally take part in in situ simulated pediatric resuscitation scenarios, as part of a team, at their institution.

STUDY PROCEDURES

Pre-Baseline Visit (online) A. Online survey (REDCap), up to 4 weeks prior to training, online questionnaires - self-report by individual providers. Time: 20-30 minutes.

Baseline Visit B. In situ simulations, team of providers participates in 2 simulated pediatric resuscitation scenarios conducted in ED. Time: 1 - 1.5 hours C. Online training module (intervention or control), individual providers will complete independently, a subset of participants present for in situ study visit will complete online training module individually between simulation sessions. Those not present for in situ study visit will complete online training module on their own. Time: 1 hour D. Post training in situ simulations, team of providers participates in 2 simulated pediatric resuscitation scenarios conducted in ED. Time: 1 - 1.5 hours Follow-up Phase (online) E. Online survey (REDCap), up to 6 weeks after online training module, online questionnaires - self-report by individual providers. Time: 20-30 minutes

STATISTICAL CONSIDERATIONS

The primary endpoint is at the provider level: pre- to post-training changes in individual providers' self-rated confidence in providing FCC in pediatric resuscitation. Investigators will also examine pre- to post-training changes in self-reported use of FCC skills in practice.

The secondary endpoint is at the site level: pre- to post-training changes in team performance of FCC, as measured by the presence and quality of family-centered care behaviors exhibited during video-recorded simulated pediatric resuscitation scenarios. Team performance measures of technical and non-technical resuscitative care skills will also be examined as a balancing measure to this endpoint.

Sample Size and Power Investigators will attempt to enroll all available providers meeting inclusion criteria at each participating ED, and estimate that approximately 300 individual participants will be enrolled, averaging 40-50 participants from each general ED site. Power analysis is based on our analyses for the primary endpoint. A sample size of 300 individuals (~150 per group) provides 80% power to detect a between-group effect size as small as .24 between groups in post-training scores, using ANCOVA.

Efficacy Analyses To evaluate the primary outcome, Investigators will examine scores on self-report surveys completed by participants before and after training. Investigators will calculate pre- to post-training change scores for individual providers, and summarize these for the total sample and by treatment group. Investigators will examine training effects on participant outcomes (self-rated confidence in providing FCC) by means of analysis of covariance (ANCOVA). In each ANCOVA, study condition will be the grouping factor and the corresponding pre-training score for the outcome measure will be included as a covariate. ANCOVA allows us to examine the potential impact of key co-variates that may vary by group despite random assignment to condition. Investigators will also estimate effect sizes for each group for pre- to post-training change in self-rated confidence in FCC skills. Investigators will then conduct parallel analyses for pre- to post-training changes in self-rated use and intentions to use FCC skills in practice with pediatric patients.

To evaluate the secondary outcome, Investigators will rate team performance based on review of video-recorded simulated pediatric resuscitations conducted before and after training. Investigators will calculate each participating site's pre- to post-intervention change in global ratings for each domain in specific aspect of FCC performance (FCC Assessment Tool), averaged across simulations and teams at that site. Investigators will also assess pre- to post-training changes in patient/scenario-specific resuscitative care (e.g., time to important interventions, success in interventions, guideline-consistent care) and in team performance (i.e. crew resource management, or CRM) using validated team performance measures (CPT and BAT). This balancing measure will allow investigators to confirm that any observed improvements in FCC do not come at the cost of poorer medical care.

Additional analyses To better understand training effects, Investigators will conduct exploratory subgroup analyses within high- and low-resource ED settings. Investigators will also conduct exploratory analyses to understand the potential impact of participation in simulated practice on clinicians' technical and non-technical resuscitation skills. Investigators will describe baseline and follow-up scores on confidence measures in these areas, and examine pre- to post changes for the subset of participants who take part in the simulation scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18 years and up.
* Healthcare providers at one of the six to eight general ED sites taking part in resuscitations as part of their usual work-related duties

Exclusion Criteria:

* Not applicable - there are no specific exclusion criteria as all providers who take part in resuscitations as part of their usual work-related duties are presumed to be capable to take part in simulation and able to read in English at the level required to complete online training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Pre- to post-training changes in individual providers' self-rated confidence in providing FCC in pediatric resuscitation | Pre-training survey up to 4 weeks prior to training, Post-training survey up to 6 weeks after training
  Pre-training to post-training change in scores on the adapted Family Presence Self-Confidence Scale (FPSCS). The FPSCS is a 29-item scale assessing health care providers' confidence in assisting patients and family members during a resuscitation, and in continuing to provide consistent high quality care while family members are present. It is on 1 to 5 scale, with 1 = not at all confident, 3 = somewhat confident, and 5 = very confident. The FPSCS total score has a potential range of 29 to 145, with higher score indicating greater confidence.
Pre- to post-training changes in self-reported use of FCC skills in practice | Pre-training survey up to 4 weeks prior to training, Post-training survey up to 6 weeks after training
  Pre-training survey up to 4 weeks prior to training, Post-training survey up to 6 weeks after training. The Use of FCC Practices survey is a 29 item questionnaire assessing for past practice of FCC skills (pre-survey) and intention to use those skills in the future (post-survey), via items adapted from the FPSCS measure described above. Responses are on a 1 to 7 scale, with 1 = never did this and 7 = did this every time. The Use of FCC Practices total score has a potential range of 29 to 203, with higher scores indicating greater use of, or intention to use, family-centered care skills in practice.

SECONDARY OUTCOMES:
Pre- to post-training changes in team performance of FCC | In situ simulations conducted immediately before and after training.
  Based on video review, expert raters (blinded) will use the FCC Assessment Tool to independently rate the quality of team performance of family-centered care during each simulation.

OTHER OUTCOMES:
Pre- to post-training changes in resuscitative care | In situ simulations conducted immediately before and after training.
  Based on video review, expert raters (blinded) will use the Clinical Performance Tool to independently rate the quality of resuscitation care during each simulation.
Pre- to post-training changes in resuscitative care and in teamwork / team performance | In situ simulations conducted immediately before and after training.
  Based on video review, expert raters (blinded) will use the Behavior Assessment Tool to independently rate the quality of teamwork / performance during each simulation.

CONTACTS AND LOCATIONS:
Overall Officials: Sage Myers, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Nancy Kassam-Adams, PhD, Principal Investigator — Children's Hospital of Philadelphia; Marc Auerbach, MD, FAAP, MSc, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale School of Medicine, New Haven, Connecticut
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No